CLINICAL TRIAL: NCT05315856
Title: Different Significance of Reactogenicity in Immunogenicity and Inflammatory Response by New COVID-19 Vaccine Platforms: BNT162b2 mRNA Versus ChAdOx1 nCoV19 Vaccine
Brief Title: Reactogenicity, Immunogenicity and Inflammatory Response by New COVID-19 Vaccine Platforms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Ajou University School of Medicine (Other); Hallym University Kangnam Sacred Heart Hospital (Other); Korean Center for Disease Control and Prevention (Other Government)
Responsible Party: Principal Investigator, Joon Young Song, Principal Investigator, Korea University Guro Hospital
Other Study IDs: 2021GR0099
Record Dates: First submitted 2022-03-29; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: COVID-19 Vaccination; Inflammation; Vaccine Immune Response; Vaccine Adverse Reaction
Keywords: reactogenicity; immunogenicity
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples Without DNA — blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- ChAdOx1 vaccine group: AstraZeneca vaccine (chimpanzee adenovirus-vectored vaccine, 0.5 mL [5 × 1010 viral particles] per dose)
  Interventions: Biological: either BNT162b2 or ChAdOx1 vaccine
- BNT162b2 vaccine group: Pfizer-BioNTech vaccine (mRNA vaccine; 0.3 mL [30 μg] per dose)
  Interventions: Biological: either BNT162b2 or ChAdOx1 vaccine

INTERVENTIONS:
Biological: either BNT162b2 or ChAdOx1 vaccine — Either BNT162b2 or ChAdOx1 was assigned to each participant by the Korean governmental policy, not allowing personal choice. Sixty participants were vaccinated with two doses of the ChAdOx1 (AstraZeneca) at 12-week intervals, and the remaining sixty were immunized with the BNT162b2 (Pfizer-BioNTech) vaccine at 3-week interval.

SUMMARY:
Analysis of humoral antibody and cytokine kinetics after vaccination with either BNT162b2 or ChAdOx1 nCoV-19 vaccine and factors influencing the vaccine immunogenicity

DETAILED DESCRIPTION:
There is a different aspect of reactogenicity between BNT162b2 and ChAdOx1 nCoV-19 vaccine. Both new platform vaccines were concerned if they would elicit more significant local or systemic reactogenicity compared to the conventional vaccines. Previous studies had reported that immune cells such as mast cells and macrophages are activated just after vaccination, and release proinflammatory cytokines such as interleukin (IL)-6 and tumor necrosis factor (TNF)-α. The post-vaccination kinetics of inflammatory cytokines would be variable by each vaccine platform, and might be associated with reactogenicity. It is an interesting issue to be investigated whether the reactogenicity following newly developed BNT162b2 and ChAdOx1 would be associated with immunogenicity and inflammatory response or not. To better clarify these uncertainties, we evaluated the change of antibody response between BNT162b2 and ChAdOx1 over three months post-vaccination, in relation to the kinetics of inflammatory cytokines and reactogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers who provide the informed consent after either BNT162b2 or ChAdOx1 vaccination
* healthy adults without underlying medical condition

Exclusion Criteria:

* Volunteers who had ever infected with SARS-CoV2 were excluded.

Ages: 19 Years to 59 Years | Sex: All
Age Groups: Adult
Study Population: Healthy young adults between the ages of 19 and 55 years who were willing to receive either BNT162b2 or ChAdOx1 were enrolled in the study and provided written informed consent
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Immunoglobulin G (IgG) anti-S antibodies | At 3 weeks after the first-dose vaccination (T1)
  measured using the Elecsys® Anti-SARS-CoV-2 S assay (Roche, Rotkreuz, Switzerland)
Immunoglobulin G (IgG) anti-S antibodies | At 3 weeks after the second-dose vaccination (T2)
  measured using the Elecsys® Anti-SARS-CoV-2 S assay (Roche, Rotkreuz, Switzerland)
Neutralizing antibodies | At 3 weeks after the first-dose vaccination (T1)
  Reduction in plaque count of 50% (PRNT50) was calculated for the median neutralizing titer (ND50) using the Spearman-Karber formula
Neutralizing antibodies | At 3 weeks after the second-dose vaccination (T2)
  Reduction in plaque count of 50% (PRNT50) was calculated for the median neutralizing titer (ND50) using the Spearman-Karber formula
IL-6, TNF-α, and IL-1ß | At 3 days after the first dose
  measured by flexible customized bead-based multiplex panels for Luminex assays (Human Premixed Multi-Analyte Kit, R&D Systems Inc., Minneapolis, MN, USA).
IL-6, TNF-α, and IL-1ß | At 3 days after the second-dose
  measured by flexible customized bead-based multiplex panels for Luminex assays (Human Premixed Multi-Analyte Kit, R&D Systems Inc., Minneapolis, MN, USA).
reactogenicity after vaccination | Until post-vaccination day 7
  Local erythema/swelling was regarded as positive sign if larger than 2.5 cm in diameter. Systemic adverse events were graded as follows: grade 0, no systemic adverse event; grade 1, any adverse event that did not interfere with activity; grade 2, any adverse event that interfered with daily activity. Fever was classified as grade 1 (from 37.5℃ to 38.4℃) and grade 2 (>38.5℃). Systemic adverse events were classified into two ways: (i) the highest level of severity of any adverse event reported by the participants and (ii) with or without specific adverse event.

SECONDARY OUTCOMES:
The correlation between humoral immune response and reactogenicity after vaccination | The correlation between reactogenicity after the first dose and immunogenicity at T1 (3 weeks after dose 1 prior to dose 2) and T2 (3 weeks after dose 2);the correlation between reactogenicity after vaccine dose 2 and immunogenicity at T2
  The correlation between humoral immune response and reactogenicity after vaccination
The correlation between cytokine response and reactogenicity after vaccination | At 3 days after each dose
  The correlation between cytokine response and reactogenicity after vaccination
Long-term immunogenicity: Immunoglobulin G (IgG) anti-S antibodies | At 3 months after the second vaccination (T3)
  measured using the Elecsys® Anti-SARS-CoV-2 S assay (Roche, Rotkreuz, Switzerland)

CONTACTS AND LOCATIONS:
Overall Officials: Joon Young Song, MD, Study Chair — Korea University Guro Hospital; Jung Yeon Heo, MD, Principal Investigator — Ajou University School of Medicine; Yu Bin Seo, MD, Principal Investigator — Hallym University Kangnam Sacred Heart Hospital
Locations (3):
- South Korea (3):
  - Ajou University School of Medicine, Suwon, Gyeonggi-do
  - Kangnam Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided
We will make a decision after discussion with the staff of other hospitals. We will share data on adverse events and immunogenicity.